CLINICAL TRIAL: NCT04690270
Title: Effects of Serotonin Receptor Agonism on Blood Glucose Lowering: Proof of Concept in Humans
Brief Title: Sumatriptan and Glucose
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Rajna Golubic, MD, PhD, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A095470; 277675 (Other: IRAS)
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Overweight
Keywords: type 1 diabetes; type 2 diabetes; glucose homeostasis; insulin secretion; insulin sensitivity; serotonin agonism
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sumatriptan 100 mg (Experimental): Given the cross-over design all participants will receive both sumatriptan (100 mg, single dose) and placebo in a random order.
  Interventions: Drug: Sumatriptan 100 mg
- Placebo (Placebo Comparator): Given the cross-over design all participants will receive both sumatriptan (100 mg, single dose) and placebo in a random order.
  Interventions: Drug: Sumatriptan 100 mg

INTERVENTIONS:
Drug: Sumatriptan 100 mg — Single dose Sumatriptan 100 mg
  Other Names: Example of a brand name for sumatriptan: Migratan

SUMMARY:
The purpose of this study is to establish the proof of concept for a brain serotonin pathway controlling blood glucose control in humans. We will examine whether activation of serotonin receptors by a single dose of sumatriptan (a drug used for the treatment of migraine) can lead to short term changes in blood glucose homeostasis. Thus far, this has been shown only in animal models but no study in humans has directly investigated this research question.

Briefly, in this study we will give a single dose of sumatriptan (100 mg) to each participant in a small sample (10 to 12) of overweight or obese, otherwise healthy humans. It will take place in the Translational Research Facility which is embedded in the Cambridge University Hospitals NHS Foundation Trust. The research staff have extensive experience and expertise in the procedures which will be used. The study will involve a screening visit and 2 subsequent visits at which sumatriptan/placebo will be taken and the glucose metabolism will be assessed using a Botnia clamp (3h procedure involving insulin and glucose infusions given intravenously with frequent blood sampling to assess insulin secretion and sensitivity). There will be about 60 days between screening visit and the last visit. The entire study (including the recruitment and data analysis) is expected to complete in about 12 months.

If sumatriptan alters glucose control, this might support future testing in disease models i.e. people with type 1 diabetes (T1D) and/or type 2 diabetes (T2D). Ultimately, if successful, either sumatriptan could be repurposed and/or other drugs from this group (triptans) could be developed for diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Being able to provide a written informed consent
2. Age between 18 and 65 years
3. Body Mass Index (BMI) ≥25 kg/m2 and <30 kg/m2 for non-Asian individuals and BMI≥23 kg/m2 and <25 kg/m2 for Asian individuals according to the BMI classification by the World Health Organization (WHO)
4. HbA1C<48 mmol/mol at screening
5. Subject must not use any regular prescribed medications (this excludes simple analgesia used as needed)
6. Subject must not use any over the counter supplements targeting metabolism
7. Subject must not have any acute or chronic disease which in the opinion of the investigator may affect the study outcome
8. Subject must not be a current smoker
9. No history of substance abuse or excess alcohol consumption (>14 units/week)
10. Women of childbearing age must have a negative pregnancy test at screening and must not be breastfeeding
11. Women of childbearing age who are sexually active with a male partner must use highly effective contraceptive methods

Exclusion Criteria:

1. Use of any regular medications
2. Use of illicit drugs
3. Use of any over the counter supplements affecting metabolism
4. Diagnosis of any acute / chronic disease
5. Current smoking or excess alcohol consumption (>14 units/week)
6. Current pregnancy or lactation
7. Abnormal findings on physical exam or routine blood tests at screening (full blood count, urea and electrolytes, HbA1C, liver function tests)
8. Concurrent participation in another trial with an investigational product
9. History of anaphylaxis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-04 (Estimated); Primary Completion 2021-06-25 (Estimated); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 1 to 4 weeks
  Change in M-value from the hyperinsulinaemic euglycaemic clamp from visit 2 to visit 3 between sumatriptan and placebo
Insulin secretion | 1 to 4 weeks
  Change in first phase insulin response from the intravenous glucose tolerance test from visit 2 to visit 3 between sumatriptan and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mark Evans, Study Chair — Institute of Metabolic Science, Hills Road, CB2 0QQ, Cambridge, UK
Locations (1):
- Rajna Golubic, Cambridge, Cambridgeshire, United Kingdom